CLINICAL TRIAL: NCT03428256
Title: A Randomised Controlled Comparison of Effectiveness of Facemask Preoxygenation and Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) in Bariatric Patients Undergoing General Anaesthesia
Brief Title: Pre-oxygenation Methods in Bariatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17SM3844
Record Dates: First submitted 2017-11-27; First posted 2018-02-09 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Anesthesia; Bariatric Surgery Candidate
Keywords: Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-oxygenation with a standard anaesthetic face mask (Active Comparator): Pre-oxygenation delivered in the standard way; 3 minutes, Fraction of inspired oxygen (FiO2) 1.0, 8 vital capacity breaths in the last minute
  Interventions: Device: Standard anaesthetic face mask
- Pre-oxygenation using Optiflow and THRIVE technique (Experimental): Pre-oxygenation delivered via nasal high flow humidified oxygen (Optiflow) and THRIVE technique. Gradually increased to 70 litres/minute, mouth closed, 8 vital capacity breaths in the last minute
  Interventions: Device: Optiflow and THRIVE technique

INTERVENTIONS:
Device: Optiflow and THRIVE technique — Nasal high flow humidified oxygen
  Arms: Pre-oxygenation using Optiflow and THRIVE technique
Device: Standard anaesthetic face mask — Oxygen delivery via an anaesthetic facemask
  Arms: Pre-oxygenation with a standard anaesthetic face mask

SUMMARY:
The purpose of the study is to compare effectiveness of different methods of achieving pre-oxygenation in bariatric patients. The investigators intend to compare facemask pre-oxygenation with a high-flow humidified nasal oxygen.

The primary outcome measure of interest is time to desaturation to 92% or 18 minutes of apnoea.

DETAILED DESCRIPTION:
General anaesthesia involves giving patients anaesthetic and muscle relaxant medications to allow transition to sleep and airway relaxation to permit laryngoscopy, respectively. During laryngoscopy, a breathing tube is placed to 'secure' the airway. There is therefore a length of time from administration of these medications to when the breathing tube is placed, when the patient is not breathing and the airway is not secured. This time is known as apnoea time. In a patient who is not breathing, blood oxygen levels fall to dangerously-low levels, within 1-2 minutes. In order to prevent this, patients breathe 100% oxygen before induction of anaesthesia as part of a process known as pre-oxygenation. There are different ways of delivering pre-oxygenation, but the common aim is to increase the oxygen reservoir within the lungs to give the anaesthetist more time to place the breathing tube. With good pre-oxygenation, apnoea times of up to 7 minutes are possible.

Apnoea time is a potentially hazardous period during induction of anaesthesia and it is particularly so in patients with severe obesity. On the one hand, obesity makes the upper airway anatomy difficult, and on the other hand, lung collapse (atelectasis) caused by abdominal contents compressing the base of the lungs reduces the amount of oxygen available within the lungs. Apnoea time can be as short of 30 seconds. Identifying the most effective method of pre-oxygenating bariatric patients can therefore significantly improve the safety of delivering general anaesthesia to these patients.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent.
* Undergoing general anaesthesia .
* Between the ages of 18 and 80 years.
* Body mass index (BMI) greater than 40 Kgm-2.

Exclusion Criteria:

* Unable to give informed consent.
* Significant cardiac history which is defined as current angina, myocardial infarction <12 months before the date of the procedure.
* Significant peripheral vascular disease defined as claudication on minimal exertion or Ankle-Brachial index of <0.7, a stroke or a transient ischaemic attack <12 months before the procedure.
* Presence of significant heart-valve disease or congestive heart failure.
* Significant lower respiratory disease including brittle asthma; chronic obstructive pulmonary disease (GOLD stages 3 or 4).
* Strong predictors of both difficult intubation and difficult facemask ventilation on anaesthetic airway assessment.
* Patient with American Society of Anesthesiologists (ASA) grade of 4 for any reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Following the induction of general anaesthesia and muscle relaxation, the time (minutes and seconds) to peripheral oxygen saturations (SpO2) of 92%. Comparing pre-oxygenation with standard face mask oxygen or THRIVE technique. | Eighteen (18) minutes maximum
  Pre-oxygenation is delivered either by a standard anaesthetic face mask or the THRIVE technique. General anaesthesia is induced and muscle relaxation is given. The time for the peripheral oxygen saturations (SpO2) to fall to 92% is recorded. When this occurs the trial is stopped and the patient is intubated.
  If 18 minutes is reached before SpO2 = 92% then the trial is stopped.

SECONDARY OUTCOMES:
The correlation between Oxygen Reserve Index (ORI) and pre-oxygenation with either a standard anaesthetic face mask or the THRIVE technique. | Eighteen (18) minutes maximum
  The investigators will simultaneously record the ORI. The ORI readings will then be correlated with the SpO2 and arterial oxygen content.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Cousins, FRCA FFICM, Principal Investigator — Imperial College Healthcare
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schutzer-Weissmann J, Wojcikiewicz T, Karmali A, Lukosiute A, Sun R, Kanji R, Ahmed AR, Purkayastha S, Brett SJ, Cousins J. Apnoeic oxygenation in morbid obesity: a randomised controlled trial comparing facemask and high-flow nasal oxygen delivery. Br J Anaesth. 2023 Jan;130(1):103-110. doi: 10.1016/j.bja.2021.12.011. Epub 2022 Jan 11. PMID 35027169